CLINICAL TRIAL: NCT04006171
Title: C Type Natriuretic Peptide and Polycystic Ovary Syndrome
Brief Title: Comparison of Serum C Type Natriuretic Peptide Levels Between Polycystic Ovary Syndrome Patients and Healthy Women
Acronym: CNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Ali Cenk, Medical Doctor, assistant professor, Near East University, Turkey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CNP
Record Dates: First submitted 2019-06-29; First posted 2019-07-05 (Actual); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Polycystic Ovary Syndrome; c Type Natriuretic Peptide; Menstrual Irregularity; Hyperandrogenism
Keywords: c type natriuretic peptide; polycystic ovary syndrome; menstrual cycle
MeSH Terms: conditions — Polycystic Ovary Syndrome; Menstruation Disturbances; Hyperandrogenism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- women with polycystic ovary syndrome (Active Comparator): 36 patients with PCOS
  Interventions: Diagnostic Test: C type natriuretic peptide
- Healthy women of reproductive age (Active Comparator): 30 patients with regular normal menstrual cycle
  Interventions: Diagnostic Test: C type natriuretic peptide

INTERVENTIONS:
Diagnostic Test: C type natriuretic peptide — Serum level of CNP in PCOS and healthy women

SUMMARY:
Recent studies have shown that C natriuretic peptide is produced from granulosa cells, increasing cumulative guanosine monophosphate (cGMP) production by affecting cumulus cells through natriuretic peptide receptors. It is suggested that produced cGMP maintains the transport of oocytes via the gap junctions and leads to a continuous increase in cyclic adenosine monophosphate (cAMP) levels in the oocyte. An important role of increased internal cAMP levels in the oocyte is shown to suppress meiotic progression.

Deoxyribonucleic acid studies in animals have shown that expression of the natriuretic peptide precursor increases during the periovulatory period and shows that this increase decreases rapidly after luteinizing hormone / human chorionic gonadotropin (hCG) stimulation.Human studies have shown that after ovulation induction, the CNP level in follicular fluid decreases following ovulatory dose of hCG.Polycystic ovary syndrome (PCOS) is the most common endocrine disease in the reproductive period, characterized by hyperandrogenism, oligo-anovulation, and polycystic ovarian morphology on ultrasonography, and in an animal study investigating the relationship between CNP and PCOS, serum CNP levels were increased in polycystic ovary syndrome.CNP serum level is thought to show differences between healthy women and women with polycystic ovary syndrome.

DETAILED DESCRIPTION:
In this prospective study, a total of 60 patients are planed to be included. PCOS group will be consisted of 30 women and control group will include 30 healthy women with regular menstruation aged between 18-40 years old. PCOS diagnosis will be made according to Rotterdam criteria.

Age and body mass index of all participants will be recorded. BMI will be calculated by dividing weight by height in square meters. Then morning fasting venous blood samples will be taken from the patients between 2nd-5th day of menstruation for both groups. All blood samples will be centrifuged on the day of collection. Sera will be aliquoted into 1.5 mL Eppendorf (Eppendorf, Milano, Italy) tubes, and will be kept at -80°C until the day of CNP test. For the PCOS patients describing oligo/anovulation, after excluding pregnancy, progesterone withdrawal bleeding will be created and then the patients will be evaluated. Serum levels of LH, FSH, estradiol, thyroid stimulating hormone (TSH), prolactin (PRL), androstenedione, dehydroepiandrosterone sulfate (DHEAS), total testosterone, free testosterone, sex hormone binding globulin (SHBG), total cholesterol (TC), triglyceride (TG), high density lipoprotein (HDL), low density lipoprotein (LDL), glucose and insulin levels will be analyzed. For insulin sensitivity, homeostatic model of insulin resistance (HOMA-IR) will be used and it will be calculated by the formula: HOMA-IR ¼ fasting blood glucose (mg/dL)fasting insulin (mIU/mL)/405. Free androgen index will be calculated by the formula 100x (Total testosteron/SHBG).

Serum CNP levels of the patients will be analyzed by an enzyme-linked immunosorbent (ELISA) assay for human C-type natriuretic peptide in accordance with the manufacturer's instructions (SEA721Hu, ELISA Kit for Human C-Type Natriuretic Peptide, Wuhan USCN Business Co., Ltd., Cloud-Clone Corp., CCC, USA).

Data will be analyzed using Statistical Packege for Social Sciences software (SPSS v15, SPSS Inc, Chicago, IL, USA). Independent t-test will be used to compare the parameters with normal distribution. Parameters that don't fulfill the parametric test assumptions will be compared using Mann-Whitney U test. Correlation of CNP with other parameters will be analyzed using Spearman's rank correlation test. Receiver operating characteristic (ROC) curve will be used to evaluate diagnostic sensitivity and specificity of CNP for PCOS. P values less than 0.05 will be regarded as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* PCOS defined according to Rotterdam criteria
* Healthy normal menstruating women

Exclusion Criteria:

* Diabetes mellitus
* Cardiavascular disease
* Renal disease
* Any drug usage
* Smoking
* Pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 90 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Özay, Principal Investigator — Near East University
Locations (1):
- Near East University Faculty of Medicine, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang M, Su YQ, Sugiura K, Xia G, Eppig JJ. Granulosa cell ligand NPPC and its receptor NPR2 maintain meiotic arrest in mouse oocytes. Science. 2010 Oct 15;330(6002):366-9. doi: 10.1126/science.1193573. PMID 20947764
- [Background] Norris RP, Ratzan WJ, Freudzon M, Mehlmann LM, Krall J, Movsesian MA, Wang H, Ke H, Nikolaev VO, Jaffe LA. Cyclic GMP from the surrounding somatic cells regulates cyclic AMP and meiosis in the mouse oocyte. Development. 2009 Jun;136(11):1869-78. doi: 10.1242/dev.035238. PMID 19429786
- [Background] Vaccari S, Weeks JL 2nd, Hsieh M, Menniti FS, Conti M. Cyclic GMP signaling is involved in the luteinizing hormone-dependent meiotic maturation of mouse oocytes. Biol Reprod. 2009 Sep;81(3):595-604. doi: 10.1095/biolreprod.109.077768. Epub 2009 May 27. PMID 19474061
- [Background] Tsafriri A, Chun SY, Zhang R, Hsueh AJ, Conti M. Oocyte maturation involves compartmentalization and opposing changes of cAMP levels in follicular somatic and germ cells: studies using selective phosphodiesterase inhibitors. Dev Biol. 1996 Sep 15;178(2):393-402. doi: 10.1006/dbio.1996.0226. PMID 8812137
- [Background] Thomas RE, Armstrong DT, Gilchrist RB. Differential effects of specific phosphodiesterase isoenzyme inhibitors on bovine oocyte meiotic maturation. Dev Biol. 2002 Apr 15;244(2):215-25. doi: 10.1006/dbio.2002.0609. PMID 11944932
- [Background] Nogueira D, Albano C, Adriaenssens T, Cortvrindt R, Bourgain C, Devroey P, Smitz J. Human oocytes reversibly arrested in prophase I by phosphodiesterase type 3 inhibitor in vitro. Biol Reprod. 2003 Sep;69(3):1042-52. doi: 10.1095/biolreprod.103.015982. Epub 2003 May 28. PMID 12773402
- [Background] Lee KB, Zhang M, Sugiura K, Wigglesworth K, Uliasz T, Jaffe LA, Eppig JJ. Hormonal coordination of natriuretic peptide type C and natriuretic peptide receptor 3 expression in mouse granulosa cells. Biol Reprod. 2013 Feb 21;88(2):42. doi: 10.1095/biolreprod.112.104810. Print 2013 Feb. PMID 23255339
- [Background] Hiradate Y, Hoshino Y, Tanemura K, Sato E. C-type natriuretic peptide inhibits porcine oocyte meiotic resumption. Zygote. 2014 Aug;22(3):372-7. doi: 10.1017/S0967199412000615. Epub 2013 Jan 18. PMID 23331536
- [Background] Kawamura K, Cheng Y, Kawamura N, Takae S, Okada A, Kawagoe Y, Mulders S, Terada Y, Hsueh AJ. Pre-ovulatory LH/hCG surge decreases C-type natriuretic peptide secretion by ovarian granulosa cells to promote meiotic resumption of pre-ovulatory oocytes. Hum Reprod. 2011 Nov;26(11):3094-101. doi: 10.1093/humrep/der282. Epub 2011 Aug 23. PMID 21865234
- [Background] Wang X, Wang H, Liu W, Zhang Z, Zhang Y, Zhang W, Chen Z, Xia G, Wang C. High level of C-type natriuretic peptide induced by hyperandrogen-mediated anovulation in polycystic ovary syndrome mice. Clin Sci (Lond). 2018 Apr 6;132(7):759-776. doi: 10.1042/CS20171394. Print 2018 Apr 16. PMID 29535265
- [Background] Reis AM, Honorato-Sampaio K. C-type natriuretic peptide: a link between hyperandrogenism and anovulation in a mouse model of polycystic ovary syndrome. Clin Sci (Lond). 2018 May 8;132(9):905-908. doi: 10.1042/CS20171491. Print 2018 May 16. PMID 29739821
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome. Fertil Steril. 2004 Jan;81(1):19-25. doi: 10.1016/j.fertnstert.2003.10.004. PMID 14711538
- [Derived] Ozay AC, Ozay OE, Edebal OH. Role of C-type natriuretic peptide in polycystic ovary syndrome. Int J Gynaecol Obstet. 2023 May;161(2):601-606. doi: 10.1002/ijgo.14568. Epub 2022 Nov 25. PMID 36373234

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were recruited from Near East University Hospital, Department of Obstetrics and Gynecology.
Pre-assignment Details: For the last 6 months, patients with drug use that may affect menstruation like oral contraceptives, patients with cardiac or renal disease and therefore drug use, patients with hypertension hystory, history of ovarian surgery, current pregnancy, hyperprolactinemia, thyroid disease, congenital adrenal hyperplasia.
Period: Overall Study
Arm/Group | Women With Polycystic Ovary Syndrome | Healthy Women of Reproductive Age
Started | 48 | 42
Completed | 36 | 30
Not Completed | 12 | 12
Not completed — Withdrawal by Subject | 8 | 7
Not completed — missing serum samples | 2 | 2
Not completed — insufficient sample volume | 2 | 3

BASELINE CHARACTERISTICS:
Population: 36 PCOS patient according to Rotterdam criterias and 30 healthy control women
Groups:
- Total: Total of all reporting groups
Arm/Group | Women With Polycystic Ovary Syndrome | Healthy Women of Reproductive Age | Total
Number analyzed (Participants) | 36 | 30 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 30 | 66
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 22 [21 to 24.8] | 24 [21.8 to 25] | 23 [21 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 30 | 66
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Cypriot | 36 | 30 | 66
Region of Enrollment [Number; unit: participants]
  Cyprus | 36 | 30 | 66
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.20 (4.26) | 21.17 (1.88) | 22.28 (3.52)

OUTCOME MEASURES:

1. Primary Outcome: Serum CNP Levels of PCOS and Healthy Participants
Description: The comparison of serum levels of C type natriuretic peptide among PCOS and healthy women
Time Frame: Second or Third Day of Menstruation
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Women With Polycystic Ovary Syndrome | Healthy Women of Reproductive Age
Number analyzed (Participants) | 36 | 30
pg/ml | 110 [90.9 to 182] | 57 [43.3 to 151.3]
Statistical Analysis 1: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p = 0.004, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Roc Curve of CNP
Description: We made a cut off value estimation for the diagnosis of PCOS by serum CNP levels using Receiver operator characteristics. The ROC curve incorporates both sensitivity (true positive rate) and specificity (true negative rate) providing a single assessment incorporating both measures. The higher the total area under the curve, the greater the predictive power of the CNP for diagnosing PCOS
Time Frame: Second or Third Day of Menstruation
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- All Participants: all participants of the study
Arm/Group | All Participants
Number analyzed (Participants) | 66
probability | 0.706 [0.574 to 0.838]
Statistical Analysis 1: Comparison: All Participants; Test type: Other; p = 0.004, Roc curve

3. Secondary Outcome: Comparison of FSH and LH of PCOS and Healthy Women
Description: Serum FSH and LH of PCOS and healthy women were compared
Time Frame: Second or Third Day of Menstruation
Population: FSH and LH should be evaluated during menstruation time period ( day 3)
Measure: Median (Inter-Quartile Range); unit: mIU/mL
Arm/Group | Women With Polycystic Ovary Syndrome | Healthy Women of Reproductive Age
Number analyzed (Participants) | 36 | 30
mIU/mL
  Follicle Stimulating Hormone | 4.7 [3.95 to 5.7] | 4.97 [4.55 to 6.06]
  Luteinizing Hormone | 4.23 [3.21 to 6.34] | 5.36 [3 to 6.89]
Statistical Analysis 1: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p = 0.171, Wilcoxon (Mann-Whitney) — p value for FSH; for FSH
Statistical Analysis 2: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p = 0.176, Wilcoxon (Mann-Whitney) — p value for LH; for LH

4. Secondary Outcome: Serum Estradiol Levels of PCOS and Healthy Women
Description: Serum Estradiol levels of PCOS and Healthy Women were compared
Time Frame: Second or Third Day of Menstruation
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Women With Polycystic Ovary Syndrome | Healthy Women of Reproductive Age
Number analyzed (Participants) | 36 | 30
pg/mL | 31 [23.5 to 45] | 36.5 [25 to 47.3]
Statistical Analysis 1: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p = 0.306, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Serum Tiroid Stimulating Hormone of PCOS and Healthy Women
Description: serum tiroid stimulating hormone of PCOS and healthy women were compared
Time Frame: Second or Third Day of Menstruation
Measure: Median (Inter-Quartile Range); unit: mIU/L
Arm/Group | Women With Polycystic Ovary Syndrome | Healthy Women of Reproductive Age
Number analyzed (Participants) | 36 | 30
mIU/L | 1.61 [1.14 to 2.15] | 1.47 [1.28 to 1.94]
Statistical Analysis 1: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p = 0.795, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Serum Prolactin Levels of PCOS and Healthy Women
Description: serum prolactin levels of PCOS and healthy women were compared
Time Frame: Second or Third Day of Menstruation
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Women With Polycystic Ovary Syndrome | Healthy Women of Reproductive Age
Number analyzed (Participants) | 36 | 30
ng/mL | 17.21 (6.65) | 16.80 (6.26)
Statistical Analysis 1: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p = 0.852, t-test, 2 sided

7. Secondary Outcome: Serum Androstenedione Levels of PCOS and Healthy Women
Description: Serum Androstenedione Levels of PCOS and Healthy Women were compared
Time Frame: Second or Third Day of Menstruation
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Women With Polycystic Ovary Syndrome | Healthy Women of Reproductive Age
Number analyzed (Participants) | 36 | 30
ng/dL | 148.89 (52.38) | 84.66 (11.56)
Statistical Analysis 1: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p < 0.001, t-test, 2 sided

8. Secondary Outcome: Serum Dehydroepiandrosterone Sulfate (DHEAS) Levels of PCOS and Healthy Women
Description: Serum dehydroepiandrosterone sulfate (DHEAS) Levels of PCOS and Healthy Women were compared
Time Frame: Second or Third Day of Menstruation
Measure: Median (Inter-Quartile Range); unit: µg/dL
Arm/Group | Women With Polycystic Ovary Syndrome | Healthy Women of Reproductive Age
Number analyzed (Participants) | 36 | 30
µg/dL | 304.55 [224.85 to 411.20] | 299.95 [213.8 to 356.3]
Statistical Analysis 1: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p = 0.277, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Serum Total Testosterone Levels of PCOS and Healthy Women
Description: Serum Total Testosterone Levels of PCOS and Healthy Women were compared
Time Frame: Second or Third Day of Menstruation
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Women With Polycystic Ovary Syndrome | Healthy Women of Reproductive Age
Number analyzed (Participants) | 36 | 30
nmol/L | 1.38 (0.48) | 0.92 (0.36)
Statistical Analysis 1: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p = 0.006, t-test, 2 sided

10. Secondary Outcome: Serum Free Testosterone Levels of PCOS and Healthy Women
Description: Serum Free Testosterone Levels of PCOS and Healthy Women were compared
Time Frame: Second or Third Day of Menstruation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Women With Polycystic Ovary Syndrome | Healthy Women of Reproductive Age
Number analyzed (Participants) | 36 | 30
pg/mL | 1.71 (0.64) | 1.12 (0.30)
Statistical Analysis 1: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p < 0.001, t-test, 2 sided

11. Secondary Outcome: Serum Sex Hormone Binding Globulin Levels of PCOS and Healthy Women
Description: Serum Sex Hormone Binding Globulin Levels of PCOS and Healthy Women were compared
Time Frame: Second or Third Day of Menstruation
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | Women With Polycystic Ovary Syndrome | Healthy Women of Reproductive Age
Number analyzed (Participants) | 36 | 30
nmol/L | 30.4 [26.8 to 53.8] | 59.4 [46.6 to 78.1]
Statistical Analysis 1: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p = 0.014, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Free Androgen Index of Participants
Description: Free androgen index of participants were compared. It was calculated with the formula 100XTotal testosterone/Sex hormone binding globulin
Time Frame: Second or Third Day of Menstruation
Measure: Mean (Standard Deviation); unit: % of T testosterone per SHBG
Arm/Group | Women With Polycystic Ovary Syndrome | Healthy Women of Reproductive Age
Number analyzed (Participants) | 36 | 30
% of T testosterone per SHBG | 4.39 (2.58) | 1.55 (0.89)
Statistical Analysis 1: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p < 0.001, t-test, 2 sided

13. Secondary Outcome: Serum Glucose, Total Cholesterol and Triglycerides Levels of Participants
Description: Serum glucose, total cholesterol and triglycerides levels of participants were compared
Time Frame: Second or third day of menstruation and morning fasting
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Women With Polycystic Ovary Syndrome | Healthy Women of Reproductive Age
Number analyzed (Participants) | 36 | 30
mg/dL
  Total cholesterol | 164 [154.3 to 185] | 171 [146 to 189]
  triglycerides | 78 [63.8 to 107.8] | 77 [60 to 90]
  Glucose | 88.5 [83.3 to 97.8] | 89 [82.3 to 94.3]
Statistical Analysis 1: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p = 0.947, Wilcoxon (Mann-Whitney) — for serum glucose; for serum glucose
Statistical Analysis 2: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p = 0.906, Wilcoxon (Mann-Whitney) — for total cholesterol; for total cholesterol
Statistical Analysis 3: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p = 0.428, Wilcoxon (Mann-Whitney) — for triglycerides; for triglycerides

14. Secondary Outcome: High Density Lipoprotein and Low Density Lipoprotein Levels of Participants
Description: High density lipoprotein and low density lipoprotein levels of participants were compared
Time Frame: Second or Third Day of Menstruation-morning fasting
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Women With Polycystic Ovary Syndrome | Healthy Women of Reproductive Age
Number analyzed (Participants) | 36 | 30
mg/dL
  High density lipoprotein | 53.82 (11.06) | 62.15 (19.48)
  Low density lipoprotein | 98.50 (23.61) | 92.92 (23.56)
Statistical Analysis 1: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p = 0.114, t-test, 2 sided — for high density lipoprotein
Statistical Analysis 2: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p = 0.504, Wilcoxon (Mann-Whitney) — for low density lipoprotein; for low density lipoprotein

15. Secondary Outcome: Serum Insulin Levels of Participants
Description: Serum Insulin Levels of Participants were compared
Time Frame: Second or Third Day of Menstruation-morning fasting
Measure: Median (Inter-Quartile Range); unit: mU/L
Arm/Group | Women With Polycystic Ovary Syndrome | Healthy Women of Reproductive Age
Number analyzed (Participants) | 36 | 30
mU/L | 7.10 [4.9 to 10] | 7.10 [5.75 to 8]
Statistical Analysis 1: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p = 0.713, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Homeostatic Model Assessment of Insulin Resistance of Participants
Description: homeostatic model assessment of insulin resistance of participants were compared. The calculation was made with formula Glucose X Insulin/405.
Time Frame: Second or Third Day of Menstruation-morning fasting
Measure: Median (Inter-Quartile Range); unit: HOMA-IR Index
Arm/Group | Women With Polycystic Ovary Syndrome | Healthy Women of Reproductive Age
Number analyzed (Participants) | 36 | 30
HOMA-IR Index | 1.50 [1.05 to 2.15] | 1.45 [1.33 to 1.88]
Statistical Analysis 1: Comparison: Women With Polycystic Ovary Syndrome vs Healthy Women of Reproductive Age; Test type: Other; p = 0.886, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were not assessed.
Description: Adverse events were not assessed.
Arm/Group | Women With Polycystic Ovary Syndrome | Healthy Women of Reproductive Age
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The limitation of our study was the relatively small number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT04006171/Prot_SAP_000.pdf